CLINICAL TRIAL: NCT03791424
Title: Changes of Skin Resistance After Midazolam and After the End of Anaesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Jiri Malek, Assoc. Prfo. Jiri Malek, CSc., Charles University, Czech Republic
Allocation: Non-Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: Oxytocin01
Record Dates: First submitted 2018-09-17; First posted 2019-01-02 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2018-12

CONDITIONS: Anesthesia
Keywords: sedation; midazolam; skin resistance; measurements
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Intervention Model Description: Multimeter DM 3900 was used for measurements of SR. The device was approved for use in humans by the Department of Medical Biophysics and Informatics of the 3rd Medical Faculty of Charles University. Observer's Assessment of Alertness and Sedation scale was used as a standard tool for measurements of sedation level at the same intervals as measurements of SR. 10 min. rest break was given to participants in order that they adapt to the test situation. The rest value of SR was noticed and next all patients were administered placebo first and after 5 min period midazolam 2 mg i.v. After next 5 minutes patients were administered standard general anaesthesia with propofol, oxygen, nitrous oxide 60 % and isoflurane 1 MAC via laryngeal mask and sufentanil as needed. Changes in skin resistance were measured again immediately after stop of volatile anaesthetics till eye opening and verbal contact.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Placebo of the same volume and colour as active substance
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Midazolam (Experimental): Midazolam 2 mg was administered 5 min. after placebo and 5 min. before inducton to general anaesthesia IV.
  Interventions: Drug: Midazolam
- Control (Placebo Comparator): Normal saline 5 ml was administered 10 min. after insertion of intravenous cannula IV..
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Midazolam — Administering premedication with sedative drug to relieve anxiety
  Other Names: Sedation

SUMMARY:
It has been described that sympathetic activity, measured as changes in electrical skin resistance (SR), may be used to assess the adequacy of general anaesthesia. Our prospective study investigated how far measurements of skin resistance can help determine level of sedation. The secondary aim was to investigate if changes in skin resistance can be used for assessing recovery from anaesthesia.

DETAILED DESCRIPTION:
Introduction Before anaesthesia, benzodiazepines are routinely used to reduce anxiety before anaesthesia and surgery. Usually anxiolysis is preferable to sedation, which may interfere with recovery after short procedures. Unfortunately, although anxiolytic sedatives are widely used in clinical practice, the methodology for assessing treatment effect of these compounds has not been well developed. Psychologic tests like the Hamilton Anxiety Rating Scale (HARS), the Wang Anxiety Rating Scale (WARS), or Zung Self-Rating Anxiety Scale (SAS) were used to assess changes in anxiety were developed for measuring effect of long-term therapy and are rather cumbersome and difficult to use in routine anaesthetic praxis.

More commonly used test in clinical perioperative use are the Ramsay sedation scale (RSS), the Richmond Agitation-Sedation Scale (RASS) and the Observer's Assessment of Alertness and Sedation scale (OAASS), but they focus mainly on level of sedation and not the level of anxiolysis. There are several reports demonstrating that there is a correlation between level of anxiety and changes in skin resistance.

Changes of skin resistance (SI) were first used in criminology in 1897 and in 1921 the method was used in criminology by August Larson together with changes of heart rate, respiratory rate and blood pressure for construction of polygraph. This method was many times validated and polygraph is still used as a "lie detector". More recently sever studies appeared demonstrating correlation between changes of skin resistance and sedation grade, bispectral index, reaction to stimulation, pain and motor activity.

The present double-blinded study was designed to refine methodology for objective evaluating effect of sedative and anxiolytic agents. The primary aim of our study was to examine if of changes in skin resistance after placebo pre-screening can be used for objective assessment of an anxiolytic effect of drugs compared to commonly used subjective scales like Ramsay sedation scale (RSS), or The Richmond Agitation-Sedation Scale (RASS) and Observer's Assessment of Alertness and Sedation scale(OAASS). The secondary aim was to evaluate if changes of skin resistance can be used for assessing recovery from anaesthesia.

Patients The study was performed in adult patients scheduled for knee arthroscopy or minor plastic surgery under general anaesthesia. Consent was obtained the day before surgery during pre-anaesthetic visit. Exclusion criteria were previous history of taking drugs affecting mental functions, history of psychic illness, implanted electrical device, know allergy to benzodiazepines, myasthenia gravis, ASA classification ASA 3 and more. All patients consented not to use any medication for sedation or anxiety, opioid analgesics, ethanol and illicit drugs 24 hours before surgery. Patients were instructed that they will be administered by a random order first sedative agent or placebo and will be observed for their level of sedation.

Measurements After arrival at the operating theatre, and venepuncture two standard AgCl ECG electrodes (Medico Electrodes International ltd.) size 32 mm x 52 mm (27x35) were attached to the palm side of the second and third finger of the non-dominating hand. Multimeter DM 3900 (Mastech) was used for measurements of SR. The device was controlled and approved for use in humans by the Department of Medical Biophysics and Informatics of the 3rd Medical Faculty of Charles University.

Observer's Assessment of Alertness and Sedation (OAAS) scale was used as a standard tool for measurements of sedation level at the same intervals as measurements of SR. The person providing OAAS assessment was blinded to the order of midazolam and placebo injection and only the anaesthetist administering both injections knew the order of drugs.

Data recording Ten min. rest break was given to participants in order that they adapt to the test situation. The rest value of SR was noticed and next all patients were administered placebo first and after 5 min period midazolam 2 mg i.v. After next 5 minutes patients were administered standard general anaesthesia with propofol, oxygen, nitrous oxide 60 % and isoflurane 1 MAC via laryngeal mask and sufentanil as needed. Monitoring was standard for this type of surgery (ECG, non-invasive blood pressure - NIBP, capnography and pulse oximetry). SR and OASS were recorded again after stop of volatile anaesthetic agent till opening eyes of the patient and obtaining verbal contact.

Statistical analysis SR values before placebo administration, 5 minutes after placebo, 5 minutes after midazolam, 5 min. after induction, at the end of surgery, 0 isoflurane level after anaesthesia with closed eyes and after eyes opening were recorded. Changes in SR values compared to baseline data were used for analyses by paired t-test. These relative changes enabled to compare only the course of changes independently of different absolute values. Pearson´s correlation coefficients were used to analyse relationship between OASS and SR values. P-value < 0.05 was considered statistically significant.

The primary aim of our study was to assess if SR can be used as an objective measurement of level of sedation compared to much or less subjective OAAS. OASS was chosen because scoring was originally introduced to assess sedation with benzodiazepines, which was used in our study, too. The categories were responsiveness, speech, facial expression and eye appearance and each category was originally scored in 5 dimensions. The OAAS scale was found to have a high discriminatory power for the different levels of sedation (3), but may vary between observers. There is a limited number of methods for assessment onset and intensity of sedation. Commonly used Bispectral Index Score (BIS) monitoring is not dependent on a person and is used mainly during general anaesthesia. On the other hand the authors of a large meta-analysis concluded that its use for sedation in largely unreliable.

ELIGIBILITY:
Inclusion Criteria:

* adult patients scheduled for knee arthroscopy or minor plastic surgery under general anaesthesia

Exclusion Criteria:

* previous history of taking drugs affecting mental functions, history of psychic illness, implanted electrical device, know allergy to benzodiazepines, myasthenia gravis, ASA classification ASA 3 and more. All patients consented not to use any medication for sedation or anxiety, opioid analgesics, ethanol and illicit drugs 24 hours before surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2015-06-26 (Actual); Study Completion 2015-06-26 (Actual)

PRIMARY OUTCOMES:
Changes of skin resistence (percent from base-line values measured in ohms) during sedation | 10 min. before administration and 5 min. after administration of midazolam (total 15 min.)
  Investigation how far measurements of skin resistance can help determine level of sedation induced by intravenous midazolam

SECONDARY OUTCOMES:
Changes of skin resistence (percent from base-line values and values before termination of inhalational agent administration measured in ohms) during recovery from anaesthesia | From termination of inhalational agent administration till recovery to verbal comunication (expected time max. 15 min)
  Investigation how far measurements of skin resistance can help determine level of recovery from general anaesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Jiri Malek, M.D., Principal Investigator — University Hospital Kralovske Vinohrady; Alice Kurzova, M.D., Study Chair — University Hospital Kralovske Vinohrady
Locations (1):
- University Hospital Kralovske Vinohrady, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No